CLINICAL TRIAL: NCT03949699
Title: Resistance Training to Improve Strength and Functional Trunk Stability in Adults With Paraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Hannah W Mercier, Postdoctoral Research Fellow, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015P001481
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: pre-post
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance Training (Other): . Participants will engage in strengthening exercises using a cable tower while seated. These movements will include trunk flexion and extension, diagonal trunk rotation, and lateral trunk flexion. The goal for resistance training frequency (Weeks 1-8) will be three times per week, lasting about 30-45 minutes per session including warm-up/cool-down. Performance during exercise sessions will be monitored by study staff who will progress the participant to exercises of greater intensity (increasing number of repetitions, sets, or resistance load; on an individual basis over the 8-week intervention period according to the participant's level of readiness). This progression will also be guided by a strength training protocol. Resistance intensity of each exercise will also be determined based on the initial maximal strength performing that exercise
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Participants will engage in strengthening exercises using a cable tower while seated. These movements will include trunk flexion and extension, diagonal trunk rotation, and lateral trunk flexion. The goal for resistance training frequency (Weeks 1-8) will be three times per week, lasting about 30-45 minutes per session including warm-up/cool-down, for a duration of eight weeks. Resistance intensity of each exercise will also be determined based on the initial maximal strength performing that exercise: Weeks 1-4 will be 50-60% of the baseline calculated 1 repetition maximum (RM) values; Weeks 5-8 will use resistive loads equivalent to 50-60% of Week 4 1RM calculations

SUMMARY:
The purpose of this study is to examine the effectiveness of an 8- week resistance training routine to improve functional trunk strength, muscle activation, and physical functioning in exercise in 30 adults with paraplegic SCI. This study will also examine outcomes of confidence in one's ability to avoid falling during balance challenges, and self-efficacy for participating in exercise activity.

DETAILED DESCRIPTION:
I. BACKGROUND AND SIGNIFICANCE Trunk stability and mobility are essential to engage in everyday life. In general, adults in the United State have weak "core" or trunk strength, resulting from weak abdominal and back musculature as well as weak muscles that assist in moving the trunk. After a spinal cord injury (SCI), the trunk becomes even less stable as there are fewer innervated muscles available to support trunk control and movement. In the absence of strong or innervated trunk-stabilizing muscles, adults with paraplegia may use compensatory patterns of maintaining an upright posture during balance challenges, which could lead to pain and musculoskeletal injury.

For these adults with paraplegia, dynamic seated postural control is greatly needed during wheelchair mobility, transfers, and safe performance of activities of daily living. This trunk control enables the individual to bend down, lean from side to side, and recover from these positions without fear of falling. Additionally, increasing trunk strength and posture and control may result in enhanced functional independence, with greater range of motion and ability to efficiently mobilize the upper extremities.

Evidence clearly indicates that strength and function declines in adults with chronic SCI can be mitigated by regular exercise, and the ability to stabilize the trunk has been thought to increase during upper body resistance training among adults with chronic paraplegia. Effective interventions that enhance trunk control and strength in this population are lacking, with preliminary studies including trunk strengthening as a preparatory activity for assisted ambulation. Furthermore, trunk strengthening is not addressed as a preventive intervention in rehabilitation for adults with paraplegia, though it is important to train whichever trunk muscles are available to support functional independence and safety.

The purpose of this study is to examine the effectiveness of an 8- week resistance training routine to improve functional trunk strength, muscle activation, and physical functioning in exercise in 30 adults with paraplegic SCI. This study will also examine outcomes of confidence in one's ability to avoid falling during balance challenges, and self-efficacy for participating in exercise activity. Participants will serve as their own control in this pre-post design.

II. SPECIFIC AIMS

1. To determine the effect of resistance training on functional postural strength, and muscle strength and activation among adults with paraplegia.

   Hypothesis: Participants who complete an 8-week resistance training program will score higher on measures of functional postural strength and muscle strength and activation.
2. To determine whether participation in an 8-week trunk resistance exercise program increases self-reported physical functioning during self-care, and basic and wheeled mobility.

   Hypothesis: Upon completing the resistance program, participants will report gains in physical functioning during activities of daily living.
3. To determine whether participation in an 8-week trunk resistance exercise program increases confidence in ability to maintain balance during daily activities and self-efficacy to participate in exercise activity.

Hypothesis: Upon completing the resistance program, participants will report declines in fear of falling, and gains in self-efficacy to participate in exercise activity.

V. STUDY PROCEDURES Methods of data collection: The proposed project is a randomized controlled study in which participants will complete a baseline assessment session. During the baseline session (Week 0 of the resistance training program), demographic and clinical data will be collected, including detailed health history. Further assessments will take place at 4-week and 8-week time points of the resistance training program. The assessments will take place in-person at Spaulding Hospital Cambridge (ExPD). Please see Study Assessments section for schedule of testing participants in either condition.

Based on their reported medical history participants may also be asked to provide additional medical records or may need further testing or physician clearance to determine their eligibility and the safety of their participation in this program which includes regular vigorous exercise (i.e. cardiology clearance, orthopedic evaluation, ASIA exam).These additional tests or medical visits may or may not be covered by insurance. The participant will be responsible for obtaining any additional testing or clearance and providing the program with medical records or results.

The duration of the entire study including recruitment, data analyses, and manuscript preparation is anticipated to be approximately 2-3 years.

Training Protocols

1) Resistance Training Group Participants will be provided up to a week (Week 0) of training to attain proficiency in using the resistance equipment, and to determine need for external assistance for safety or to adjust resistance levels and cables. Participants will engage in strengthening exercises using a cable tower while seated. These movements will include trunk flexion and extension, diagonal trunk rotation, and lateral trunk flexion. The goal for resistance training frequency (Weeks 1-8) will be three times per week, lasting about 30-45 minutes per session including warm-up/cool-down, for a duration of eight weeks. Performance during exercise sessions will be monitored by study staff that will progress the participant to exercises of greater intensity (increasing number of repetitions, sets, or resistance load; on an individual basis over the 8-week intervention period according to the participant's level of readiness). This progression will also be guided by a strength training protocol, as each participant indicates s/he are doing well with the exercises, are not experiencing pain, and specify a decrease in the challenge level of particular exercises. Resistance intensity of each exercise will also be determined based on the initial maximal strength performing that exercise: Weeks 1-4 will be 50-60% of the baseline calculated 1 repetition maximum (RM) values; Weeks 5-8 will use resistive loads equivalent to 50-60% of Week 4 1RM calculations; the final session during Week 8 will be used to determine final strength values (see Measurement and Testing Protocols below for further details).

There is no limit or specific requirement for training sessions that must be attended to continue participating in this protocol. Subjects will be encouraged by study staff to attend three training sessions per week. Un-reported missed training session will be followed up with a phone call to document why the training session was missed and to encourage prompt return to training sessions as soon as possible.

ELIGIBILITY:
Inclusion Criteria: To be included in the study, all subjects must be adults (>18 years of age) and:

* Be in good health (asymptomatic for acute treatable illness)
* Be able to understand, communicate with and be understood by research personnel and interpreters
* Be interested in participating and provide informed consent
* Have a SCI with residual deficits (AIS A, B, C), and from the neurological level of T2 and lower to allow at least partial use of trunk muscles
* Use a wheelchair as primary means of mobility (≥6 hours/day)

Exclusion Criteria: Participants must not be enrolled in any strengthening protocol or rehabilitation therapy for strengthening during the time of the study. Participants must not have serious comorbidities that could interfere with the ability to participate in an exercise program (musculoskeletal, cardiovascular, and neurological [other than SCI]). Specifically, participants will be excluded if they have: 1) Musculoskeletal injuries that have not healed completely, 2) Had heart surgery or are status post-myocardial infarction (MI) in the last 4 to 6 months, 3) Unstable angina, 4) Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg), 5) uncontrolled dysrhythmias, 6) Recent history of congestive heart failure that has not been evaluated and effectively treated, 7) Severe stenotic or regurgitant valvular disease, or 8) Hypertrophic cardiomyopathy.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Change in Strength | . Testing will be repeated at weeks 4 & 8. Maximum strength values established during Baseline and 4th week testing will be used to calculate the exercise workloads for the next four weeks of training
  Maximum strength: Subjects will be given a set of ten repetitions with a light weight, as a warm-up prior to testing. The weight stack will then be adjusted to a load intended to induce muscular fatigue within ten repetitions. The subject will perform as many complete repetitions as possible. Once the subject fails to perform a repetition through the complete range of motion, they will have reached fatigue, and the weight and number of repetitions will be recorded. If the number of repetitions exceeds ten, then the weight will be increased and the subject will be given a three-minute rest interval before repeating the test. A regression equation 4 will then be used to calculate maximum strength
Change in Balance | Baseline, and weeks 4 & 8
  Items from the Activity-based Balance Level Evaluation (ABLE) Sitting Balance subscale: Participants perform the following activities, which are scored according to ability and quality of movement: 1.Sitting with back unsupported but feet supported on floor or on a foot stool; 2. Modified functional reach test; 3. Seated lateral reach; 4. Pick up an object from the floor from a seated position; 5. Scooting forward in a chair; and 6. External perturbations in sitting. This measure typically takes 15 minutes to administer.

SECONDARY OUTCOMES:
Change in SCI-Functional Index (SCI-FI) | Baseline and 8 weeks
  A self-report computer-adapted test measuring difficulty performing activities in the domains of Basic Mobility, Self-Care, and Wheelchair Mobility. This measure typically takes less than 7 minutes to administer
Change in Falls Concern Scale for people with SCI (SCI-FCS) | Baseline and 8 weeks
  A questionnaire that asks respondents to rate their level of concern about the possibility of falling during 16 daily activities. Ratings are given on a 4-point Likert scale from Not at all concerned (1) to very concerned (4). This measure typically takes 5 minutes or less to complete.
Change in SCI Exercise Self-Efficacy Scale (SCI ESES) | Baseline and 8 weeks
  Participants respond to 10 items on a 4-point Likert-style scale (1-not at all true, 4-always true) that is used to determine likelihood of the respondent to engage in exercise activity. This measure typically takes less than 5 minutes to administer.